CLINICAL TRIAL: NCT03607370
Title: Timing for Rectal Surgery After ChST
Brief Title: Timing for Rectal Surgery After Chemoradiotherapy
Acronym: ST812
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center Affiliate of Vilnius University Hospital Santaros Klinikos (Other)
Responsible Party: Principal Investigator, Audrius Dulskas, Assoc. profesor, National Cancer Center Affiliate of Vilnius University Hospital Santaros Klinikos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST812
Record Dates: First submitted 2018-06-20; First posted 2018-07-31 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Chemoradiotherapy; Surgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (No Intervention): The cancer surgery is practice 8 weeks after neoadjuvant chemoradiotherapy
- Group 2 (Experimental): The cancer surgery will be performed in 12 weeks after neoadjuvant chemoradiotherapy
  Interventions: Procedure: Surgery after 12 weeks of delay after chemoradiotherapy.

INTERVENTIONS:
Procedure: Surgery after 12 weeks of delay after chemoradiotherapy. — Surgery consists oncologic resection of the rectal cancer with total excision of the mesorectum after 12 weeks of delay after the end of chemoradiotherapy.
  Arms: Group 2

SUMMARY:
The aim of this study is to determine whether greater rectal cancer downstaging and regression occurs when surgery is delayed to 12 weeks after completion of radiotherapy/chemotherapy compared to 8 weeks.

Hypothesis: Greater down-staging and tumor regression is observed when surgery is delayed to 12 weeks after completion of chemoradiotherapy compared to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Eastern Cooperative Oncology Group (ECOG) 0-1,
* American Society of Anesthesiologists' (ASA) score I-III
* Histological confirmation of adenocarcinoma of rectum
* T3 or T4 N0, T any N positive cancer on MRI, without metastasis on CT scan
* Undergoing preoperative radiotherapy/ chemotherapy
* Curative total mesorectal excision intended
* Written informed consent
* Patients undergoing preoperative radiotherapy should not be excluded

Exclusion Criteria:

* Patients with distant metastasis
* T1 or T2, N0 cancer on MRI
* Rectal cancer 12 cm above the dentate line
* Contraindications to MRI
* Patients previously treated of pelvic organ cancer
* Medical or psychiatric conditions that compromise the patients ability to give informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete pathologic response assessed by pathologist Dworak scale | 6 months
  Dworak scale assesses the response: 0. No regression; 1. Predominantly tumor with significant fibrosis and/or vasculopathy; 2. Predominantly fibrosis with scattered tumor cells (slightly recognizable histologically); 3. Only scattered tumor cells in the space of fibrosis with/without acellular mucin; 4. No vital tumor cells detectable

SECONDARY OUTCOMES:
Clinical response assessed using MRi | 8 weeks (2 months)
  Rates of clinical response to chemoradiotherapy before surgery, comparison between the two groups
Pathological response assessed by pathologist using Dworak scale | 6 months
  Dworak scale assesses the response: 0. No regression; 1. Predominantly tumor with significant fibrosis and/or vasculopathy; 2. Predominantly fibrosis with scattered tumor cells (slightly recognizable histologically); 3. Only scattered tumor cells in the space of fibrosis with/without acellular mucin; 4. No vital tumor cells detectable
Incidence of Treatment-Emergent Adverse Events as assessed by Clavien-Dindo scale | 30 days
  Rates of operative morbidity at 30 days, comparison between the two groups. Grade I Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions Allowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgetics, diuretics and electrolytes and physiotherapy. This grade also includes wound infections opened at the bedside.
  Grade II Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Blood transfusionsand total parenteral nutritionare also included. Grade III Requiring surgical, endoscopic or radiological intervention
  * IIIa Intervention not under general anesthesia
  * IIIb Intervention under general anesthesia Grade IV Life-threatening complication (including CNS complications)* requiring IC/ICU-management
  * IVa single organ dysfunction (including dialysis)
  * IVb multiorgan dysfunction
Incidence of Mortality assessed by Clavien-Dindo scale | 30 days
  Rates of operative mortality at 30 days, comparison between the two groups. Grade V Death of a patient
Total mesorectal excision (TME) quality assessed by TME completeness scale (by P.Quircke) | 8-12 weeks
  Quality of mesorectum resection assessed by TME completeness scale:
  1. Mesorectal resection (MRR)/good/complete: intact mesorectum and smooth mesorectal surface with only minor irregularities; no defects deeper than 5 mm; no coning of the specimen towards the distal margin; and smooth macro-circular resection margin (CRM) on slicing.
  2. Intramesorectal resection (IMR)/intermediate/nearly complete: intermediate bulk of the mesorectum with an irregular surface; a defect deeper than 5 mm, and no visible muscularis propria other than inserted levator; intermediate coning; intermediate irregularity of macro-CRM on slicing.
  3. Muscularis propria resection (MPR)/poor/incomplete: small bulk of the mesorectum with a very irregular surface; defect down to the muscularis propria; severe coning; severe irregularity of macro-CRM on slicing.
Distant recurrence assessed by CT scan | 5 years
  Distant recurrence rates, comparison between the two groups
Local recurrence assessed by CT scan/MRI/endoscopy | 5 years
  Local recurrence rates, comparison between the two groups
Oncological outcome - overall survival | 5 years
  Overall survival rates, comparison between the two groups
Oncological outcome - disease-free survival | 5 years
  Disease-free survival rates, comparison between the two groups
Radiotherapy skin toxicity assessed by EORTC scale | 5 years
  Radiotherapy related toxicity rates: skin reactions will be assessed using EORTC radiotherapy toxicity scale: Skin Grade 1 follicular, faint or dull erythema / epilation / dry desquamation / decreased sweating; Grade 2 tender or bright erythema, patchy moist desquamation / moderate edema; Grade 3 confluent, moist desquamation other than skin folds, pitting edema; Grade 4 - ulceration, hemorrhage, necrosis
Radiotherapy toxicity assessed by EORTC scale | 5 years
  Radiotherapy related toxicity rates: gastrointestinal reactions will be assessed using EORTC radiotherapy toxicity scale:
  Grade 1 increased frequency or change in quality of bowel habits not requiring medication / rectal discomfort not requiring analgesics; Grade 2 diarrhea requiring parasympatholytic drugs (e.g. Lomotil) / mucous discharge not necessitating sanitary pads / rectal or abdominal pain requiring analgesics; Grade 3 diarrhea requiring parenteral support / severe mucous or blood discharge necessitating sanitary pads / abdominal distention (flat plate radiograph demonstrates distended bowel loops); Grade 4 acute or subacute obstruction, fistula or perforation; GI bleeding requiring transfusion; abdominal pain or tenesmus requiring tube decompression or bowel diversion
Quality of Life assessed by Low anterior resection syndrome score | 1 year
  The Low anterior resection syndrome score (LARS) score consists of five items concerning the following: incontinence for flatus, incontinence for liquid stool, frequency of bowel movements, clustering of stools, and urgency. Each symptom of bowel dysfunction is weighed according to its impact on the quality of life. The calculated score ranges from 0 to 42, with a score of 0-20 representing no ARS, a score of 21-29 representing minor ARS, and a score of 30-42 representing major ARS.
Immune response assessed | 1 year
  We have assessed the immune response before chemoradiotherapy and 8 weeks following the treatment. IL1B, IL6, IL8, IL10, IL2R, TNF alfa are assessed and will be correlated with the response to treatment.
Urinary catheter removal timing | 3 months
  All the patients will have there urinary catheters removed on day 1. Some patients will get Urorec (adrenomimetic for prevention of urinary retention). The patients will be randomized 2:1

CONTACTS AND LOCATIONS:
Overall Officials: Audrius Dulskas, MD, PhD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Vilnius, Lithuania

REFERENCES:
- [Derived] Didrikaite G, Klimovskij M, Civilka I, Buckus B, Aukstikalnis T, Sileika E, Dulskas A. Quality of life following ileostomy takedown: single-centre, retrospective clinical trial-does closure time matter? Tech Coloproctol. 2025 Jul 30;29(1):154. doi: 10.1007/s10151-025-03196-2. PMID 40736758
- [Derived] Gricius Z, Kuliavas J, Stratilatovas E, Buckus B, Dulskas A. Early urinary catheter removal in patients undergoing rectal cancer surgery: a randomized controlled trial on silodosin versus no pharmacological treatment on urinary function in the early postoperative period. Ann Coloproctol. 2025 Jun;41(3):239-245. doi: 10.3393/ac.2024.00703.0100. Epub 2025 Jun 20. PMID 40537941